CLINICAL TRIAL: NCT06381128
Title: Detection of Coronary Arteries Anomalies by Computed Tomography Angiography in Children With Congenital Heart Disease
Brief Title: Coronary Arteries Anomalies by CT in Children With CHD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Rashed Gad, RMRGad, Assiut University
Other Study IDs: CAA by CT in children with CHD
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Congenital Defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Cardiac CT — Computed tomography angiography

SUMMARY:
Delineate coronary artery anatomy and detection of coronary anomalies in children with complex cardiac anomalies by cardiac CT-angiography before total surgical correction.

DETAILED DESCRIPTION:
Congenital heart diseases (CHD) form an important spectrum of pediatric diseases causing significant morbidity and mortality. Due to inter-related embryology of the heart and development of the coronary arteries, there is a great variability in coronary artery patterns in patients with CHD [1].

The spectrum of coronary artery anomalies ranges from benign / incidental findings to significant cardiac morbidity in infancy or increased risk of cardiac sudden death in childhood or adolescence [2]. Abnormalities can be found in the coronary artery origin, course, and size or the number of vessels. Isolated anomalies of coronary artery origins, in those without structural heart disease, had an estimated incidence of 0.7% [3]. Coronary artery anomalies have a higher incidence in children with congenital heart disease, ranging from an incidence of 5% in those with coarctation [4] to 7% in tetralogy of Fallot [5] and up to 37% in single-ventricle physiologies [6]. Identifying these anomalies has become an important part of the preoperative evaluation to avoid inadvertent injury and has been shown to be effectively diagnosed with modern CT techniques compared to surgical visualization and catheter angiography [6,7]. System of coronary artery origin and branching is of great help to surgeons who dedicate their efforts to the treatment of congenital heart disease [8].

Coronary artery imaging in children is frequently challenging due to small size, high heart rates, and motion artifacts from cardiac pulsation, respiration, and the patients themselves, which results in technical or procedural difficulties [9].

Imaging modalities for evaluating coronary arteries in children include echocardiography, conventional invasive angiography, magnetic resonance imaging (MRI), and computed tomography (CT). Transthoracic echocardiography is widely used as the primary imaging approach. However, it is impaired by its limited ability to fully characterize coronary anatomy, by poor acoustic windows, and by operator dependency [10].

Magnetic resonance imaging (MRI), also provides information on cardiac anatomy and function, allowing 3-dimensional coronary artery imaging without the use of ionizing radiation.However, it is impaired by long acquisition time requiring prolonged patient cooperation, which may not be possible in children without general anesthesia, and bylimited spatial resolution which makes coronary evaluation beyond originassessment difficult [11].

Computed tomography (CT) angiography is often the firstline diagnostic modality of choice for noninvasive imaging of the coronary arteries in both adults and children. CT is rapidly acquired and can be performed in the setting of multiple support devices. Compared with cardiac MRI and transthoracic echocardiography, CT provides excellent spatial resolution with superior visualization of the entire course of the coronary arteries [12].

Recent advances in CT technology have allowed for dramatic decreases in radiation dose while maintaining theexcellent spatial resolution that allows for detailed anatomical evaluation [13].

Coronary artery abnormalities in children may be congenital or acquired. Congenital anomalies include a complex group of disorders occurring as isolated conditions or in the spectrum of congenital heart disease.Acquired coronary anomalies are mainly secondary to Kawasaki disease or surgery when congenital heart disease repair involves coronary manipulation. Increasing evidence is supporting the role of CT in general for coronary evaluation of these patients [14,15]. The Coronary artery anomalies are grouped under four subtypes, i.e. anomalies of origin and course, intrinsic anomalies of coronaries, anomalies of termination, and anomalous anastomotic vessels [16]. Coronary artery abnormalities are more common in patients with congenital heart disease. Even when clinically irrelevant, these lesions may become important as they may affect surgical repair. Unambiguous coronary artery imaging is therefore mandatory in this situation and, especially when echocardiography is not conclusive ,CT should be employed to avoid unnecessary invasive procedures, even in the neonatal period. The most common conditions to consider in this setting include tetralogy of Fallot and (dextro-)transposition of the great arteries[17].

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 1 day to 18 years old with congenital heart disease and undergoing surgical correction.

Exclusion Criteria:

* 1-Children had isolated coronary anatomy anomalies.

  2-Children had medical coronary artery disease i.e. Kawasaki disease.

  3-Children with CHD and not candidate for surgical correction .

  4-Children with CHD with past history of cardiac surgery.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: -Children aged from 1 day to 18 years old with congenital heart disease and undergoing surgical correction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of coronary arteries anomalies by computed tomography angiography in children with congenital heart disease | Baseline
  Delineate coronary artery anatomy and detection of coronary anomalies in children with complex cardiac anomalies by cardiac CT-angiography before total surgical correction.

REFERENCES:
- [Background] Jacobs ML, Mavroudis C. Anomalies of the coronary arteries: nomenclature and classification. Cardiol Young. 2010 Dec;20 Suppl 3:15-9. doi: 10.1017/S1047951110001046. PMID 21087555
- [Background] Cheezum MK, Liberthson RR, Shah NR, Villines TC, O'Gara PT, Landzberg MJ, Blankstein R. Anomalous Aortic Origin of a Coronary Artery From the Inappropriate Sinus of Valsalva. J Am Coll Cardiol. 2017 Mar 28;69(12):1592-1608. doi: 10.1016/j.jacc.2017.01.031. PMID 28335843
- [Background] Mery CM, De Leon LE, Molossi S, Sexson-Tejtel SK, Agrawal H, Krishnamurthy R, Masand P, Qureshi AM, McKenzie ED, Fraser CD Jr. Outcomes of surgical intervention for anomalous aortic origin of a coronary artery: A large contemporary prospective cohort study. J Thorac Cardiovasc Surg. 2018 Jan;155(1):305-319.e4. doi: 10.1016/j.jtcvs.2017.08.116. Epub 2017 Sep 14. PMID 29074047
- [Background] Vastel-Amzallag C, Le Bret E, Paul JF, Lambert V, Rohnean A, El Fassy E, Sigal-Cinqualbre A. Diagnostic accuracy of dual-source multislice computed tomographic analysis for the preoperative detection of coronary artery anomalies in 100 patients with tetralogy of Fallot. J Thorac Cardiovasc Surg. 2011 Jul;142(1):120-6. doi: 10.1016/j.jtcvs.2010.11.016. Epub 2011 Feb 3. PMID 21292283
- [Background] Yu FF, Lu B, Gao Y, Hou ZH, Schoepf UJ, Spearman JV, Cao HL, Sun ML, Jiang SL. Congenital anomalies of coronary arteries in complex congenital heart disease: diagnosis and analysis with dual-source CT. J Cardiovasc Comput Tomogr. 2013 Nov-Dec;7(6):383-90. doi: 10.1016/j.jcct.2013.11.004. Epub 2013 Nov 8. PMID 24331934
- [Background] Secinaro A, Curione D, Mortensen KH, Santangelo TP, Ciancarella P, Napolitano C, Del Pasqua A, Taylor AM, Ciliberti P. Dual-source computed tomography coronary artery imaging in children. Pediatr Radiol. 2019 Dec;49(13):1823-1839. doi: 10.1007/s00247-019-04494-2. Epub 2019 Aug 22. PMID 31440884
- [Background] Frommelt P, Lopez L, Dimas VV, Eidem B, Han BK, Ko HH, Lorber R, Nii M, Printz B, Srivastava S, Valente AM, Cohen MS. Recommendations for Multimodality Assessment of Congenital Coronary Anomalies: A Guide from the American Society of Echocardiography: Developed in Collaboration with the Society for Cardiovascular Angiography and Interventions, Japanese Society of Echocardiography, and Society for Cardiovascular Magnetic Resonance. J Am Soc Echocardiogr. 2020 Mar;33(3):259-294. doi: 10.1016/j.echo.2019.10.011. No abstract available. PMID 32143778
- [Background] Goo HW. Coronary artery imaging in children. Korean J Radiol. 2015 Mar-Apr;16(2):239-50. doi: 10.3348/kjr.2015.16.2.239. Epub 2015 Feb 27. PMID 25741188
- [Background] Lederlin M, Thambo JB, Latrabe V, Corneloup O, Cochet H, Montaudon M, Laurent F. Coronary imaging techniques with emphasis on CT and MRI. Pediatr Radiol. 2011 Dec;41(12):1516-25. doi: 10.1007/s00247-011-2222-0. Epub 2011 Nov 30. PMID 22127683
- [Background] Hazekamp M. Coronary Anatomy in Congenital Heart Disease: The Important Contributions of Professor Dr. Adriana Gittenberger-de Groot. J Cardiovasc Dev Dis. 2021 Mar 9;8(3):27. doi: 10.3390/jcdd8030027. PMID 33803117
- [Background] Freire G, Miller MS. Echocardiographic evaluation of coronary arteries in congenital heart disease. Cardiol Young. 2015 Dec;25(8):1504-11. doi: 10.1017/S1047951115002000. PMID 26675597
- [Background] Malone LJ, Morin CE, Browne LP. Coronary computed tomography angiography in children. Pediatr Radiol. 2022 Dec;52(13):2498-2509. doi: 10.1007/s00247-021-05209-2. Epub 2021 Nov 4. PMID 34734316
- [Background] Ezzeldin DA, Hafez MS, Mansour A. Multidetector computed tomography for patients with congenital heart disease: a multi-center registry from Africa and Middle East; patients' characteristics and procedural safety. Egypt Heart J. 2021 Oct 16;73(1):90. doi: 10.1186/s43044-021-00217-x. PMID 34655343
- [Background] Zhang LJ, Zhou CS, Wang Y, Jin Z, Yu W, Zhang Z, Zhang B, Fang X, Cui X, Li K, Huang W, Zheng L, Ji XM, Hoffman C, Schoepf UJ, Lu GM. Prevalence and types of coronary to pulmonary artery fistula in a Chinese population at dual-source CT coronary angiography. Acta Radiol. 2014 Nov;55(9):1031-9. doi: 10.1177/0284185113512299. Epub 2013 Nov 26. PMID 24280135
- [Background] Chao BT, Wang XM, Wu LB, Chen J, Cheng ZP, Wu DW, Duan YH. Diagnostic value of dual-source CT in Kawasaki disease. Chin Med J (Engl). 2010 Mar 20;123(6):670-4. PMID 20368084
- [Background] Kashyap JR, Kumar S, Reddy S, Rao K R, Sehrawat O, Kashyap R, Kansal M, Reddy H, Kadiyala V, Uppal L. Prevalence and Pattern of Congenital Coronary Artery Anomalies in Patients Undergoing Coronary Angiography at a Tertiary Care Hospital of Northern India. Cureus. 2021 Apr 10;13(4):e14399. doi: 10.7759/cureus.14399. PMID 33981512
- [Background] Han BK, Rigsby CK, Hlavacek A, Leipsic J, Nicol ED, Siegel MJ, Bardo D, Abbara S, Ghoshhajra B, Lesser JR, Raman S, Crean AM; Society of Cardiovascular Computed Tomography; Society of Pediatric Radiology; North American Society of Cardiac Imaging. Computed Tomography Imaging in Patients with Congenital Heart Disease Part I: Rationale and Utility. An Expert Consensus Document of the Society of Cardiovascular Computed Tomography (SCCT): Endorsed by the Society of Pediatric Radiology (SPR) and the North American Society of Cardiac Imaging (NASCI). J Cardiovasc Comput Tomogr. 2015 Nov-Dec;9(6):475-92. doi: 10.1016/j.jcct.2015.07.004. Epub 2015 Jul 23. PMID 26272851